CLINICAL TRIAL: NCT01381237
Title: Full Title Interactive Computer Game Exercise Regime, Effects on Balance Impairment in Frail Community-Dwelling Older Adults. A Randomized Controlled Trial
Brief Title: Effects of Game-based Balance Exercise for Older Adults With Fall History
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Dr. Tony Szturm, Associate Professor, Dept. of Physical Therapy, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2007-047
Record Dates: First submitted 2011-06-20; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2007-03

CONDITIONS: Mobility Limitation
Keywords: Balance; Postural; Rehabilitation; Therapy; computer-assisted; Video Games; Center of Pressure
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: game-based balance exercises — 16 sessions, scheduled two per week, each lasting 45 minutes.

SUMMARY:
Due to the many problems associated with reduced balance and mobility, providing an effective and engaging rehabilitation regimen is essential to progress recovery from impairments and to help prevent further degradation of motor skills. The purpose was to examine effects of physical therapy based on the task-oriented approach delivered in an engaging, interactive video game paradigm. The intervention focused on performing targeted dynamic tasks, which included reactive balance controls and environmental interaction. Thirty community dwelling and ambulatory older adults attending the Day hospital for balance and mobility limitation treatment participated in this study. Participants were randomly assigned to either a control group or experimental group. The control group received the typical rehabilitation program provided at the Day Hospital, consisting of strengthening and balance exercises. The experimental group received a program of dynamic balance exercises coupled to video game play, using a centre of pressure (COP) position signal as the computer mouse. The tasks were performed while standing on a fixed floor surface with progression to a compliant sponge pad. Each group received 16 sessions, scheduled two per week, each lasting 45 minutes. Balance performance measures and spatial-temporal gait variables were obtained pre- and post-treatment Findings demonstrated significant improvements for both groups in balance performance scores post-treatment, and change scores were significantly greater in the experimental compared to control group. No significant treatment effect was observed in either group for the spatial-temporal gait variables. In conclusion dynamic balance exercises on fixed and compliant sponge surfaces were feasibly coupled to interactive game-based exercise. This in turn resulted in a greater improvement in dynamic standing balance control compared to the typical exercise program. However there was no transfer of effect to gait function.

Key Words: Balance, Postural; Rehabilitation; Therapy, computer-assisted; Video Games; Center of Pressure.

ELIGIBILITY:
Inclusion Criteria:

* age: 65-85 years
* Mini-Mental State Examination (MMSE) score > 24
* English-speaking with the ability to understand the nature of the study and provide informed consent
* independent in ambulatory functions, with or without an assistive device (cane or walker).

Exclusion Criteria:

* any medical condition or disability that prevented participation in an exercise program.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Standing Balance | 5 weeks
  timed performance and ordinal scales

SECONDARY OUTCOMES:
Gait speed | 5 weeks
Spatial-temporal gait variables | 5 weeks
  distance and time

CONTACTS AND LOCATIONS:
Overall Officials: Tony Szturm, BSc(PT), PhD, Principal Investigator — University of Manitoba
Locations (1):
- Riverview Health Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Szturm T, Betker AL, Moussavi Z, Desai A, Goodman V. Effects of an interactive computer game exercise regimen on balance impairment in frail community-dwelling older adults: a randomized controlled trial. Phys Ther. 2011 Oct;91(10):1449-62. doi: 10.2522/ptj.20090205. Epub 2011 Jul 28. PMID 21799138